CLINICAL TRIAL: NCT05504005
Title: Clinical Validation of Multi-channel Microspatial Offset Raman Scattering Spectroscopy (mμSORS) for Noninvasive Blood Glucose Detection
Brief Title: Clinical Validation of mμSORS for Noninvasive Blood Glucose Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Photonic View Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCEMD2022002
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus; Medical Device
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Validation of mμSORS for Noninvasive Blood Glucose Detection (Experimental): Enrolled subjects will perform oral glucose tolerance test. A measurement session of blood glucose consists of plasma sample and a measurement by mμSORS will be conducted synchronously.
  Interventions: Device: Multi-channel Microspatial Offset Raman Scattering Spectroscopy (mμSORS) for Noninvasive Blood Glucose Detection

INTERVENTIONS:
Device: Multi-channel Microspatial Offset Raman Scattering Spectroscopy (mμSORS) for Noninvasive Blood Glucose Detection — Blood glucose of participants were measured by venous plasma and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS). The two measurements were collected synchronously and analyzed.

SUMMARY:
This is a single-center, open-label, prospective study. Blood glucose was measured at different time points during oral glucose tolerance testing in healthy subjects and patients with type 2 diabetes mellitus, using both venous plasma and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS). Venous plasma glucose was set as gold standard.The two measurements were collected synchronously so as to calculate the mean absolute relative difference (MARD) and the consensus error grid (CEG). Accuracy of non-invasive blood glucose testing by mμSORS will be validated. MARD for two measurement methods in different blood glucose ranges and the effect of mμSORS on safety in the patient such as adverse events will also be assessed.

DETAILED DESCRIPTION:
In order to clinically verify the accuracy and safety of non-invasive blood glucose measurement by the mμSORS technology, and to construct a model, this study will conduct oral glucose tolerance tests on healthy subjects and patients with type 2 diabetes at different time points during the OGTT. There will be 12 points as follows: 0-min and post glucose-load 10-min，30-min，60-min，90-min，120-min，150-min，180-min，210-min，240-min，270-min， and 300-min.

ELIGIBILITY:
Inclusion Criteria for healthy subjects:

* Male or female.
* Aged between 30 and 60 years.
* Fasting blood glucose (FPG) < 6.1 mmol/L and glycated hemoglobin (HbA1c) < 5.7% during the screening period.
* There are no scars, obvious pigmentation and other factors that interfere with the detection of the palm skin to be tested.
* Confirmed as healthy based on the results of physical examination, medical history, vital signs and clinical laboratory tests.
* Fully understand the nature, significance, possible benefits, possible inconveniences or potential risks of this research, and should also understand the research procedures, be willing to complete the entire research process, and provide written consent form.

Inclusion Criteria for patients with type 2 diabetes:

* Male or female，previously diagnosed type 2 diabetes.
* Aged between 30 and 60 years.
* Fasting plasma glucose ≥ 6.1 and < 13.3 mmol/L.
* There are no scars, obvious pigmentation and other factors that interfere with the detection of the palm skin to be tested.
* Fully understand the nature, significance, possible benefits, possible inconveniences or potential risks of this research, and should also understand the research procedures, be willing to complete the entire research process, and provide written consent form.

Exclusion Criteria for healthy subjects:

* Any history of serious clinical diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry or metabolic abnormality, or any other disease that can interfere with the test results, which the investigator considers significant.
* Alcohol dependency or drug abuse.
* Those who have participated in clinical trials of other drugs within 3 months before screening (since the last visit of the previous trial).
* Pregnancy or lactation period.
* Difficulty in venous blood collection or fainting of needles or blood.
* Other circumstances that the investigator considers inappropriate to participate in the study.

Exclusion Criteria for patients with type 2 diabetes:

* Type 1 diabetes, monogenic mutant diabetes, pancreatic damage, or secondary diabetes of other causes should be excluded.
* Severe structural heart disease, such as congenital heart disease, rheumatic heart disease, hypertrophic or dilated cardiomyopathy, chronic congestive heart failure (NYHA≥III); acute myocardial infarction within 12 months before enrollment; history of severe liver or kidney dysfunction (eGFR < 60 ml/min/1.73m2 calculated by MDRD formula at screening period); and mental disorders, etc.
* With a history of acute complications of diabetes within 3 months before enrollment; or severe diabetes-related complications.
* Alcohol dependency or drug abuse.
* Those who have participated in clinical trials of other drugs within 3 months before screening (since the last visit of the previous trial).
* Pregnancy or lactation period.
* Difficulty in venous blood collection or fainting of needles or blood.
* Other circumstances that the investigator considers inappropriate to participate in the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 35 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Mean absolute relative deviation (MARD) of venous plasma glucose and glucose values measured by mμSORS at each time point of OGTT. | 2 months
  Glucose will be measured using both intravenous sampling (plasma) and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS) detection synchronously.
Consensus Error Grid (CEG) for venous plasma glucose and glucose values measured by mμSORS at each time point of OGTT. | 2 months
  Glucose will be measured using both intravenous sampling (plasma) and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS) detection synchronously.

SECONDARY OUTCOMES:
MARD for two measurement methods in different blood glucose ranges. | 2 months
  Plasma glucose ranges 3.9-10.0 mmol/L, <3.9 mmol/L and >10.0 mmol/L.
Incidence of Treatment-Emergent Adverse Events | 2 months
  Safety in the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Wang, Dr., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China